CLINICAL TRIAL: NCT02875340
Title: A Phase II Study to Assess the Efficacy, Safety and Tolerability of VAL401 in the Treatment of Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) After Failure of at Least One Prior Chemotherapeutic Regimen
Brief Title: A Study of VAL401 in the Treatment of Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ValiSeek Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAL401-001
Record Dates: First submitted 2016-08-15; First posted 2016-08-23 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VAL401 treatment (Experimental): Patients received VAL401 oral formulation once daily according to their level of tolerance (2 mg - 10 mg).
  Interventions: Drug: VAL401

INTERVENTIONS:
Drug: VAL401 — Risperidone formulated into a liquid lipid filled capsule
  Other Names: Risperidone lipid formulation

SUMMARY:
The objectives of this study are to assess the safety, tolerability, pharmacokinetics and efficacy of VAL401 in the treatment of patients with locally advanced or metastatic non-small cell lung adenocarcinoma.

DETAILED DESCRIPTION:
This is a Phase II, open label study to assess the efficacy, safety and tolerability of VAL401 in the treatment of patients with locally advanced or metastatic non-small cell lung adenocarcinoma after failure of at least one prior chemotherapeutic regimen. Eligible patients will be enrolled as a single cohort and treated with VAL401, given as oral capsules. VAL401 is a formulation of Risperidone (active pharmaceutical ingredient) in a liquid lipid filled capsule.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of Stage IIIB or Stage IV adenocarcinoma of the lung. Patients with mixed histology will be eligible if adenocarcinoma is the predominant histology.
* Measurable disease according to RECIST version 1.1.
* Prior chemotherapy for relapsed or metastatic non small cell lung cancer.
* Life expectancy of at least 3 months.
* Negative human chorionic gonadotropin (hCG) test in women of childbearing potential (defined as women ≤ 50 years of age or history of amenorrhea for ≤ 12 months prior to study screening). Sexually active male and female patients of childbearing potential must agree to use an effective method of birth control e.g. barrier methods with spermicides, oral or parenteral contraceptives and/or intrauterine devices, during the entire duration of the study and for 1 month after the final administration of VAL401. Note that female patients may be surgically sterile (with appropriate documentation in the patient's medical records).
* Ability to give written, informed consent prior to any study-specific screening procedures with the understanding that the consent may be withdrawn by the patient at any time without prejudice.
* Patient is capable of understanding the protocol requirements, is willing and able to comply with the study protocol procedures, and has signed the informed consent document.

Exclusion Criteria:

* Radiotherapy or surgery (other than biopsy) within 4 weeks prior to Cycle 1 Day 1.
* Any chemotherapy regimens (including investigational agents) with delayed toxicity with 6 weeks of Cycle 1 Day 1, or received any chemotherapy regimens given continuously or on a weekly basis which have limited potential for delayed toxicity within 2 weeks prior to Cycle 1 Day 1. Palliative treatment regimens, and other concomitant drugs regimens are permitted with stable toxicity, and recording of all concomitant medications (including herbal).
* Pregnant or lactating female patients.
* Active hepatitis B or C or other active liver disease (other than malignancy).
* Any active, clinically significant, viral, bacterial, or systemic fungal infection within 2 weeks prior to Cycle 1 Day 1; other than cytomegalovirus which may be present providing any required concomitant anti-viral treatment is recorded appropriately.
* Known human immunodeficiency virus positivity.
* History of clinically significant cardiac condition, including ischemic cardiac event, myocardial infarction or unstable cardiac disease with 3 months prior to Cycle 1 Day 1.
* Active brain metastases (defined as stable for <4 weeks and/or symptomatic and/or requiring treatment with anticonvulsants or steroids and/or leptomeningeal disease).
* Any known contraindications to Risperidone or patients who would not be eligible to receive the treatment as defined in the Special Warnings and Precautions section of the local label for Risperidone.
* Any medical history that in the Investigator's opinion would jeopardise compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data will be made available on primary and secondary endpoints within 12 months of database lock.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 31 October 2016 - 19 June 2017
Period: Overall Study
Arm/Group | VAL401 Treatment
Started | 8
Completed | 0 (No patients completed 6 months of continuous treatment)
Not Completed | 8
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | VAL401 Treatment
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 65.8 [54 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Georgia | 8
Smokers [Count of Participants; unit: Participants]
  Smokers | 0
  Ex-smokers | 4
  Never-smokers | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from screening to disease progression (or death if the patient died before progression), with progression date nominally defined as the date the patient was withdrawn from the trial, where the Principal Investigator has determined by their professional discretion the patient has symptomatic disease progression.
Time Frame: 6 months
Measure: Mean (Full Range); unit: weeks
Groups:
- VAL401 Treatment - Intention to Treat Group: Patients received VAL401 oral formulation once daily according to their level of tolerance (2 mg - 10 mg).
  This group includes all patients who completed screening, but excludes the one patient for whom the date of diagnosis is inconsistent.
- VAL401 Treatment - Per Protocol Group: Patients received VAL401 oral formulation once daily according to their level of tolerance (2 mg - 10 mg).
  This groups excludes the 2 patients received treatment for less than 10 days, as well as the patient for whom the date of diagnosis is inconsistent.
Arm/Group | VAL401 Treatment - Intention to Treat Group | VAL401 Treatment - Per Protocol Group
Number analyzed (Participants) | 7 | 5
weeks | 5.2 [0.4 to 11.6] | 7.2 [4.0 to 11.6]

2. Secondary Outcome: Patient Quality of Life During VAL401 Treatment
Description: Changes in patient quality of life measured by EORTC Health-related Quality of Life (HRQoL) assessment questionnaire QLQ-C30 (Cancer specific questionnaire).
Time Frame: 6 months
Population: Each question is scored on a scale of 1 to 4, with each patient assessed for improvement or deterioration of Quality of Life for each life category stated. The number of patients, improving, deteriorating or remaining stable for each measure is reported out of the total of 8 patients assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | VAL401 Treatment
Number analyzed (Participants) | 8
Participants
  ECOG data: Not measured | 4
  ECOG data: Status maintained | 3
  ECOG data: Status deteriorated | 1
  ECOG data: Status improved | 0
  Improvement in pain: Not measured | 2
  Improvement in pain: Status maintained | 2
  Improvement in pain: Status deteriorated | 0
  Improvement in pain: Status improved | 4
  Improvement in Insomnia: Not measured | 2
  Improvement in Insomnia: Status maintained | 3
  Improvement in Insomnia: Status deteriorated | 1
  Improvement in Insomnia: Status improved | 2
  Improvement in lack of appetite: Not measured | 2
  Improvement in lack of appetite: Status maintained | 3
  Improvement in lack of appetite: Status deteriorated | 1
  Improvement in lack of appetite: Status improved | 2
  Improvement in nausea/vomiting: Not measured | 2
  Improvement in nausea/vomiting: Status maintained | 4
  Improvement in nausea/vomiting: Status deteriorated | 0
  Improvement in nausea/vomiting: Status improved | 2
  Improvement in fatigue: Not measured | 2
  Improvement in fatigue: Status maintained | 1
  Improvement in fatigue: Status deteriorated | 2
  Improvement in fatigue: Status improved | 3
  Improvement in irritability: Not measured | 2
  Improvement in irritability: Status maintained | 2
  Improvement in irritability: Status deteriorated | 3
  Improvement in irritability: Status improved | 1
  Improvement in depression: Not measured | 2
  Improvement in depression: Status maintained | 2
  Improvement in depression: Status deteriorated | 2
  Improvement in depression: Status improved | 2
  Improvement in anxiety: Not measured | 2
  Improvement in anxiety: Status maintained | 1
  Improvement in anxiety: Status deteriorated | 3
  Improvement in anxiety: Status improved | 2
  Improvement in diarrhoea: Not measured | 2
  Improvement in diarrhoea: Status maintained | 4
  Improvement in diarrhoea: Status deteriorated | 1
  Improvement in diarrhoea: Status improved | 1

3. Secondary Outcome: Number of Participants Reporting Adverse Events and Serious Adverse Events
Description: Ongoing evaluation of Adverse Events during treatment with VAL401. Events assessed for number of patients affected, severity of event, likelihood of event being related to the drug treatment and whether the event is an expected/known side effect of Risperidone.
Time Frame: 6 months
Population: Total number of patients reporting Adverse Events or Serious Adverse Events (excluding death)
Measure: Count of Participants; unit: Participants
Arm/Group | VAL401 Treatment
Number analyzed (Participants) | 8
Participants
  Adverse Events reported: Number participants reporting events | 8
  Adverse Events reported: Number participants reporting no events | 0
  Serious Adverse Events Reported: Number participants reporting events | 1
  Serious Adverse Events Reported: Number participants reporting no events | 7

4. Secondary Outcome: Number of Patients With Disease Control
Description: Objective tumour response rates according to RECIST 1.1 for target lesions and assessed by CT:
  Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: 6 months
Population: Participants scheduled to receive scans at screening, 3 months and 6 months. 2 participants attended CT scans at 3 months, or at their final visit (if earlier).
Measure: Count of Participants; unit: Participants
Arm/Group | VAL401 Treatment
Number analyzed (Participants) | 2
Participants
  Participants receiving mid-treatment CT scan | 2
  Primary target tumour increased by 10% or less | 2
  Participants demonstrating Complete Response | 0
  Participants demonstrating Partial Response | 0
  Participants demonstrating Progressive disease | 0
  Participants demonstrating Stable Disease | 2

5. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: Assessment of Cmax in collected blood samples on Day 1 and Day 15 of Cycle 1, collected at time points: pre-dose (0h) then 10, 15, 30 minutes, 1, 2, 4, 8, 10 and 24 hours after administration of VAL401.
Time Frame: 1 Day and 2 weeks
Population: Pharmacokinetic measurements include total of Risperidone plus metabolite 9-hydroxy-Risperidone as "total actives"
  Note: 3 out of 8 patients completed PK analysis at Day 15, the remaining 5 patients did not undergo Day 15 PK analysis due to protocol deviations or early withdrawal from the trial.
Measure: Mean (Full Range); unit: ng/mL
Groups:
- VAL401 Treatment - Day 1: Patients received VAL401 oral formulation once daily according to their level of tolerance (2 mg - 10 mg)
- VAL401 Treatment - Day 15 (2 mg): Pharmacokinetic measurements taken on Day 15 of dosing on 2 mg daily dose level
- VAL401 Treatment - Day 15 (6 mg): Pharmacokinetic measurements taken on Day 15 of dosing on 6 mg daily dose level
- VAL401 Treatment - Day 15 (8 mg): Pharmacokinetic measurements taken on Day 15 of dosing on 8 mg daily dose level
Arm/Group | VAL401 Treatment - Day 1 | VAL401 Treatment - Day 15 (2 mg) | VAL401 Treatment - Day 15 (6 mg) | VAL401 Treatment - Day 15 (8 mg)
Number analyzed (Participants) | 8 | 1 | 1 | 1
ng/mL | 30.5 [13 to 65] | 20 [20 to 20] | 102 [102 to 102] | 464 [464 to 464]

6. Secondary Outcome: Trough Plasma Concentration (Cmin)
Description: Assessment of trough plasma concentration (Cmin) in collected blood samples on Day 1 and Day 15 of Cycle 1, collected at time points: pre-dose (0h) then 10, 15, 30 minutes, 1, 2, 4, 8, 10 and 24 hours after administration of VAL401.
Time Frame: 1 Day and 2 weeks
Population: Pharmacokinetic measurements include total of Risperidone plus metabolite 9-hydroxy-Risperidone as "total actives".
  Note: 3 out of 8 patients completed PK analysis at Day 15, the remaining 5 patients did not undergo Day 15 PK analysis due to protocol deviations or early withdrawal from the trial.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | VAL401 Treatment - Day 1 | VAL401 Treatment - Day 15 (2 mg) | VAL401 Treatment - Day 15 (6 mg) | VAL401 Treatment - Day 15 (8 mg)
Number analyzed (Participants) | 8 | 1 | 1 | 1
ng/mL | 10.125 [4 to 26] | 11 [11 to 11] | 35 [35 to 35] | 111 [111 to 111]

7. Secondary Outcome: Plasma VAL401 Half-life (t 1/2)
Description: Assessment of plasma half-life of VAL401 (t 1/2) in collected blood samples on Day 1 and Day 15 of Cycle 1, collected at time points: pre-dose (0h) then 10, 15, 30 minutes, 1, 2, 4, 8, 10 and 24 hours after administration of VAL401.
Time Frame: 1 Day and 2 weeks
Population: as for outcome 6
Measure: Mean (Full Range); unit: hours
Arm/Group | VAL401 Treatment - Day 1 | VAL401 Treatment - Day 15 (2 mg) | VAL401 Treatment - Day 15 (6 mg) | VAL401 Treatment - Day 15 (8 mg)
Number analyzed (Participants) | 8 | 1 | 1 | 1
hours | 9 [7 to 36] | 26 [26 to 26] | 30 [30 to 30] | 16 [16 to 16]

8. Secondary Outcome: Overall Survival
Description: Defined as the time from screening to death if the patient dies within the period that the site is open
Time Frame: 6 months
Measure: Mean (Full Range); unit: weeks
Arm/Group | VAL401 Treatment - Intention to Treat Group | VAL401 Treatment - Per Protocol Group
Number analyzed (Participants) | 7 | 5
weeks | 7.8 [0.4 to 15.3] | 10.9 [6.9 to 15.3]

ADVERSE EVENTS:
Time Frame: Adverse Event data collected from time of screening until patient final visit (up to 6 months)
Arm/Group | VAL401 Treatment
All-Cause Mortality (participants affected / at risk) | 3/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAL401 Treatment (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAL401 Treatment (N=8)
Fatigue (Social circumstances) | 6 (9)
Vertigo (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sleepiness (Social circumstances) | 2 (6)
Nervousness (Nervous system disorders) | 2 (2)
Excitement (Nervous system disorders) | 2 (2)
Agression (Nervous system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bifasicular block (Cardiac disorders) | 1 (1)
Supraventricular extrasystole (Cardiac disorders) | 1 (1)
Ventricular extrasystole (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (5)
Peripheral venous thrombosis (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Pericardial effusion (Vascular disorders) | 1 (1)
Pleural effusion (Vascular disorders) | 1 (1)
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
ALP rise (Hepatobiliary disorders) | 1 (1)
Left lower extremity edema (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study initially planned to recruit up to 20 patients, but closed recruitment at 8 patients due to operational challenges, and the limitations of data coming in, due to frailty of end stage cancer patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT02875340/Prot_SAP_000.pdf